CLINICAL TRIAL: NCT04532931
Title: Phase 2, Exploratory, Single Center, Randomized, Open Label, Adaptive Clinical Trial to Compare Safety and Efficacy of Four Different Experimental Drug Regimens to Standard of Care for the Treatment of Symptomatic Outpatients With COVID-19
Brief Title: Four Different Experimental Drug Regimens to Standard of Care for the Treatment of Symptomatic Outpatients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP-PA-COV-202
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: COVID-19; Pyramax; Pyronaridine; Artesunate; Chloroquine; Zinc; Amodiaquine; Favipiravir; Nitazoxanide; Sofosbuvir; Daclatasvir
MeSH Terms: conditions — COVID-19 | interventions — Acetaminophen; amodiaquine, artesunate drug combination; pyronaridine tetraphosphate, artesunate drug combination; favipiravir; nitazoxanide; Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Paracetamol (SOC) (Placebo Comparator): 500 mg oral tablets. Two tablets taken at 6-hour intervals as needed, in all treatment arms (in addition to any investigative treatment)
  Interventions: Drug: Paracetamol
- Artesunate-amodiaquine (ASAQ) (Experimental): Fixed dose combination tablets containing 100 mg artesunate and 270 mg amodiaquine. Participants received two tablets once daily for 3 days
  Interventions: Drug: Artesunate-amodiaquine
- Pyronaridine-artesunate (PA) (Experimental): Fixed dose combination tablets containing 180 mg pyronaridine and 60 mg artesunate, given once daily for 3 days. Participants weighing 45 to <65 kg received 3 tablets per dose, those ≥65 kg received 4 tablets per dose
  Interventions: Drug: Pyronaridine-artesunate
- Favipiravir plus nitazoxanide (FPV-NTZ) (Experimental): Free combination of favipiravir 200 mg and 400 mg tablets and nitazoxanide 500 mg tablets. Participants received favipiravir as a loading dose of 1600 mg twice daily for 1 day followed by 600 mg twice daily for 6 days, and nitazoxanide 1000 mg twice daily, with food, for 7 days
  Interventions: Drug: Favipiravir plus Nitazoxanide
- SOC plus Sofosbuvir/daclatasvir (Experimental): Fixed dose combination tablets containing 400 mg sofosbuvir and 60 mg daclatasvir. Participants received 1 tablet once daily for 7 days
  Interventions: Drug: Sofosbuvir/daclatasvir

INTERVENTIONS:
Drug: Paracetamol — SOC - 2 tablets (1000 mg) to be taken 6-hourly as needed
  Other Names: Control treatment (SoC)
  Arms: Paracetamol (SOC)
Drug: Artesunate-amodiaquine — SOC plus artesunate-amodiaquine (ASAQ) - 2 tablets (200/540 mg artesunate/amodiaquine) daily for 3 days
  Other Names: ASAQ
  Arms: Artesunate-amodiaquine (ASAQ)
Drug: Pyronaridine-artesunate — SOC plus pyronaridine-artesunate (PA) Weight 45 to <65 kg: 3 tablets (540/180 mg pyronaridine/artesunate) daily for 3 days Weight ≥65 kg: 4 tablets (720/240 mg pyronaridine/artesunate) daily for 3 days
  Other Names: PA
  Arms: Pyronaridine-artesunate (PA)
Drug: Favipiravir plus Nitazoxanide — SOC plus favipiravir plus nitazoxanide (FPV-NTZ) Favipiravir: 1600 mg 12-hourly for 1 day then 600 mg 12-hourly for 6 days Nitazoxanide: 2 tablets (1000 mg) 12-hourly for 7 days
  Other Names: FPV-NTZ
  Arms: Favipiravir plus nitazoxanide (FPV-NTZ)
Drug: Sofosbuvir/daclatasvir — SOC plus sofosbuvir/daclatasvir (SOF/DCV)
  1 tablet (400 mg/60 mg sofosbuvir/daclatasvir) daily for 7 days
  Other Names: SOF/DCV
  Arms: SOC plus Sofosbuvir/daclatasvir

SUMMARY:
This exploratory study is a randomized, single center, open label study of four different experimental treatment arms versus standard of care for the treatment of SARS-CoV-2 infection in symptomatic outpatients with mild disease at the time of enrollment.

DETAILED DESCRIPTION:
This phase 2, exploratory study will be an adaptive, randomized, open label, trial for treatment of individuals in an outpatient settings with mild SARS-CoV-2 infection. The primary outcome is focused on the evaluation of efficacy of the proposed experimental drugs in reducing upper respiratory viral shedding, defined as viral clearance (i.e., negative swab) on Day 7. Key secondary outcomes focus on other measures of viral shedding, safety evaluation, progression to LRTI (defined by resting blood oxygen saturation level [SpO2] <93% sustained for two readings two hours apart and presence of subjective dyspnoea or cough), disease severity, clinical resolution rate, and cumulative incidence of hospitalization or mortality at Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 65 years of age, inclusive, at the time of signing the informed consent.
2. Willing and able to provide informed consent.
3. Women of reproductive potential must be using a highly effective method of contraception for at least 28 days prior to enrolment and must be able and willing to continue its use throughout the duration of the study.
4. Men must agree to use condoms when engaging in heterosexual sex during the study and for the period up to 91 days after the last dose of study medication. Men who are not randomized to a treatment arm including favipiravir (or another arm identified as having teratogenic potential through semen) will no longer need to adhere to this after randomization.
5. Laboratory confirmed SARS-CoV-2 infection, and any of the following self-reported symptoms within 72 hours prior to randomization: fever or chills, cough, myalgia, sore throat, shortness of breath, or new onset of anosmia or ageusia.
6. Body weight ≥45 kg.
7. Access to reliable video conference, telephone, direct/text messaging, or other device permitting real-time, reliable information transfer.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Known hypersensitivity or specific contraindications to the use of any of the active drugs in the treatment arms, or similar compounds.
3. Signs of respiratory distress prior to randomization, including:

   * respiratory rate >24 breaths/min
   * SpO2 <95% in room air.
4. Resting pulse rate ≥120 beats/min.
5. High likelihood of hospitalization in the opinion of the attending clinician.
6. QTcF >470 msec for females, or >450 msec for males, at screening.
7. Serum potassium <3.5 mmol/L at screening.
8. History of clinically significant cardiovascular disease (including arrhythmias, QT-interval prolongation, torsades de pointes (TdP), history of coronary artery disease with graft or stent procedures/surgery, cardiac failure [class 2 or higher using the New York Heart Association functional classification]).
9. Known chronic kidney disease (Stage IV or receiving dialysis).
10. Known cirrhosis (Child-Pugh Class B or greater).
11. Known macular degeneration, or other known retinal diseases, or 4-aminoquinolone-induced visual impairment.
12. Currently receiving, or recently received (within 60 days prior to randomization) treatment with any of the drugs in the treatment arms.
13. Currently receiving, or recently received (within 30 days prior to randomization) treatment with any antimalarial drugs.
14. Currently on treatment with drugs with known arrhythmogenic potential, or those known to induce significant QT-interval prolongation or TdP, as detailed in Appendix 6.
15. Currently on treatment for tuberculosis (or on treatment with rifampicin for any other indication), or on treatment with a protease inhibitor-based antiretroviral regimen, or efavirenz, or carbamazepine.
16. Inability/unlikely to be in the study area for the duration of the 28 day follow-up period.
17. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the volunteer or the objectives of the study. The Investigator should make this determination in consideration of the volunteer's medical history.
18. Personnel (e.g. investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study.
19. Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Venter, PhD, Principal Investigator — Ezintsha, Wits Reproductive Health & HIV Institute University of the Witwatersrand
Locations (1):
- Ezintsha, Wits Reproductive Health & HIV Institute University of the Witwatersrand, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Paracetamol (SOC): Standard of care (Paracetamol): SOC - 2 tablets (1000 mg) to be taken 6-hourly as needed
- SOC Plus Artesunate-Amodiaquine: Artesunate-amodiaquine: SOC plus artesunate-amodiaquine (ASAQ) - 2 tablets (200/540 mg artesunate/amodiaquine) daily for 3 days
- SOC Plus Favipiravir Plus Nitazoxanide: Favipiravir plus Nitazoxanide: SOC plus favipiravir plus nitazoxanide (FPV-NTZ) Favipiravir: 1600 mg 12-hourly for 1 day then 600 mg 12-hourly for 6 days Nitazoxanide: 2 tablets (1000 mg) 12-hourly for 7 days
- SOC Plus Pyronaridine-Artesunate: Pyronaridine-artesunate: SOC plus pyronaridine-artesunate (PA) Weight 45 to <65 kg: 3 tablets (540/180 mg pyronaridine/artesunate) daily for 3 days Weight ≥65 kg: 4 tablets (720/240 mg pyronaridine/artesunate) daily for 3 days
Period: Overall Study
Arm/Group | Paracetamol (SOC) | SOC Plus Artesunate-Amodiaquine | SOC Plus Favipiravir Plus Nitazoxanide | SOC Plus Pyronaridine-Artesunate | SOC Plus Sofosbuvir/Daclatasvir
Started | 39 | 39 | 38 | 38 | 38
Completed | 37 | 39 | 36 | 36 | 35
Not Completed | 2 | 0 | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Paracetamol (SOC): Paracetamol (SOC)
  Standard of care (Paracetamol): SOC - 2 tablets (1000 mg) to be taken 6-hourly as needed
- ASAQ: SOC plus Artesunate-Amodiaquine
  Artesunate-amodiaquine: SOC plus artesunate-amodiaquine (ASAQ) - 2 tablets (200/540 mg artesunate/amodiaquine) daily for 3 days
- PA(Pyronaridine-Artesunate): SOC plus Pyronaridine-Artesunate
  Pyronaridine-artesunate: SOC plus pyronaridine-artesunate (PA) Weight 45 to <65 kg: 3 tablets (540/180 mg pyronaridine/artesunate) daily for 3 days Weight ≥65 kg: 4 tablets (720/240 mg pyronaridine/artesunate) daily for 3 days
- FPV-NTZ: SOC plus Favipiravir plus Nitazoxanide
  Favipiravir plus Nitazoxanide: SOC plus favipiravir plus nitazoxanide (FPV-NTZ) Favipiravir: 1600 mg 12-hourly for 1 day then 600 mg 12-hourly for 6 days Nitazoxanide: 2 tablets (1000 mg) 12-hourly for 7 days
- SOF/DCV: SOC plus Sofosbuvir/daclatasvir
  Sofosbuvir/daclatasvir: SOC plus sofosbuvir/daclatasvir (SOF/DCV)
  1 tablet (400 mg/60 mg sofosbuvir/daclatasvir) daily for 7 days
- Total: Total of all reporting groups
Arm/Group | Paracetamol (SOC) | ASAQ | PA(Pyronaridine-Artesunate) | FPV-NTZ | SOF/DCV | Total
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35 | 186
Age, Categorical [Count of Participants; unit: Participants] — Population: Percentages are based on the number participants in the mITT analysis set Participants in all investigational treatment arms received SoC in addition to the respective experimental treatment
  Participants
    <=18 years | 0 | 0 | 1 | 0 | 0 | 1
    Between 18 and 65 years | 39 | 39 | 35 | 37 | 35 | 185
    >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (9.93) | 36 (10.32) | 35.9 (11.28) | 34 (9.43) | 34.8 (10.58) | 34.9 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Percentages are based on the number participants in the mITT analysis set Participants in all investigational treatment arms received SoC in addition to the respective experimental treatment
  Participants
    Female | 24 | 25 | 20 | 15 | 15 | 99
    Male | 15 | 14 | 16 | 22 | 20 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Percentages are based on the number participants in the mITT analysis set Participants in all investigational treatment arms received SoC in addition to the respective experimental treatment
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 2 | 3 | 0 | 1 | 1 | 7
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 36 | 32 | 34 | 32 | 31 | 165
    White | 1 | 2 | 2 | 2 | 1 | 8
    More than one race | 0 | 2 | 0 | 2 | 2 | 6
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Percentages are based on the number participants in the mITT analysis set Participants in all investigational treatment arms received SoC in addition to the respective experimental treatment
  Participants
    South Africa: Black African | 36 | 32 | 34 | 32 | 31 | 165
    South Africa: Coloured | 0 | 2 | 0 | 2 | 2 | 6
    South Africa: White | 1 | 2 | 2 | 2 | 1 | 8
    South Africa: Asian or Indian | 2 | 3 | 0 | 1 | 1 | 7
    South Africa: Other | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of SARS-CoV-2 Clearance
Time Frame: Day 7
Measure: Number; unit: percentage of paticaipants
Groups:
- Arm A: Paracetamol (SOC)
  Standard of care (Paracetamol): SOC - 2 tablets (1000 mg) to be taken 6-hourly as needed
- Arm B: SOC plus Artesunate-Amodiaquine
  Artesunate-amodiaquine: SOC plus artesunate-amodiaquine (ASAQ) - 2 tablets (200/540 mg artesunate/amodiaquine) daily for 3 days
- Arm C: SOC plus Pyronaridine-Artesunate
  Pyronaridine-artesunate: SOC plus pyronaridine-artesunate (PA) Weight 45 to <65 kg: 3 tablets (540/180 mg pyronaridine/artesunate) daily for 3 days Weight ≥65 kg: 4 tablets (720/240 mg pyronaridine/artesunate) daily for 3 days
- Arm D: SOC plus Favipiravir plus Nitazoxanide
  Favipiravir plus Nitazoxanide: SOC plus favipiravir plus nitazoxanide (FPV-NTZ) Favipiravir: 1600 mg 12-hourly for 1 day then 600 mg 12-hourly for 6 days Nitazoxanide: 2 tablets (1000 mg) 12-hourly for 7 days
- Arm E: SOC plus Sofosbuvir/daclatasvir
  Sofosbuvir/daclatasvir: SOC plus sofosbuvir/daclatasvir (SOF/DCV)
  1 tablet (400 mg/60 mg sofosbuvir/daclatasvir) daily for 7 days
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
percentage of paticaipants | 34.2 | 38.5 | 30.3 | 27.0 | 23.5

2. Secondary Outcome: Incidence of SARS-CoV-2 Clearance
Time Frame: Day 3, 10, 14, 21, 28
Measure: Number; unit: percentage of paticaipants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
percentage of paticaipants
  Day 3 | 28.2 | 17.9 | 17.1 | 24.3 | 14.3
  Day 10 | 33.3 | 33.3 | 40.0 | 29.7 | 34.3
  Day 14 | 56.4 | 51.3 | 45.7 | 51.4 | 51.4
  Day 21 | 66.7 | 53.8 | 68.6 | 64.9 | 68.6
  Day 28 | 71.8 | 66.7 | 68.6 | 73.0 | 68.6

3. Secondary Outcome: Time to Clearance of Nasal SARS-CoV-2
Time Frame: Day 0, 3, 7, 10, 14, 21, 28
Measure: Median (95% Confidence Interval); unit: Time(day)
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Time(day) | 10 [7 to 14] | 7 [3 to 9] | 8.5 [3 to 14] | 14 [3 to 14] | 8.5 [3 to 14]

4. Secondary Outcome: Estimated Viral Load of SARS-CoV-2 Detected by Quantitative RT-PCR
Description: baseline and day14, Day 14 value minus baseline value
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: Log₁₀ copies/mL
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Log₁₀ copies/mL | -3.81 (2.576) | -3.35 (2.531) | -3.30 (2.283) | -3.50 (2.691) | -2.98 (2.757)

5. Secondary Outcome: Poisson Regression for Proportion of Days With Fever After Randomization
Time Frame: Day 28
Measure: Number; unit: proportion
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
proportion | 0.596 | 0.000 | 1.732 | 0.599 | 0.835

6. Secondary Outcome: Percentage of Days With Respiratory Symptoms After Randomization
Description: "Percentage of total study days in which participants experienced respiratory symptoms until day 28. Percentage calculated as (No. of days with respiratory symptoms) ÷ (No. of days observation) x 100"
Time Frame: from randomization to end of study (until day 28)
Measure: Mean (95% Confidence Interval); unit: Percentage (%)
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Percentage (%) | 35.66 [28.252 to 38.450] | 28.034 [22.134 to 30.386] | 33.469 [26.451 to 36.416] | 29.602 [23.947 to 32.937] | 35.306 [30.099 to 40.711]

7. Secondary Outcome: FLU-PRO Plus Questionnaire Scores and FLU-PRO Plus Global Additional Daily Diary Items Over the First 14 Days
Description: baseline and day 14, Day 14 value minus baseline value The FLU-PRO(inFLUenza Patient-Reported Outcome) Plus questionnaire was completed daily during the first 14 days, at Day 21 and at Day 28.
  From these items six domain scores for the body areas Nose, Throat, Eyes, Chest/Respiratory, Gastrointestinal, and Body/Systemic could be computed ranging from 0 (symptom free) to 4 (very severe symptoms).
  Total Score Range for FLU-PRO Plus
  * Score range per item: 0 (no symptoms) to 4 (very severe symptoms). A higher score indicates worse symptoms.
  * Total score calculation: The mean (average) of all item scores is used. (Minimum score: 0, Maximum score: 4)
Time Frame: 14 days
Measure: Median (Standard Deviation); unit: score
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
score | -0.750 (0.8270) | -0.750 (1.0046) | -0.750 (0.9079) | -1.250 (0.9135) | -0.750 (0.5711)

8. Secondary Outcome: Serious Adverse Events
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 38 | 36 | 36
Participants | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Adverse Events
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Participants | 0 | 0 | 0 | 1 | 1

10. Secondary Outcome: Related Adverse Events
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Participants | 0 | 11 | 12 | 21 | 10

11. Secondary Outcome: LRTI
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Participants | 0 | 0 | 2 | 0 | 1

12. Secondary Outcome: Maximum Score on WHO Ordinal Scale for Clinical Improvement During Study Participation
Time Frame: Day 28
Measure: Median (Standard Deviation); unit: score
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
score | 1 (0.5) | 0 (0.6) | 1 (0.76) | 1 (0.43) | 1 (0.81)

13. Secondary Outcome: Cumulative Incidence of Hospitalization
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Participants | 0 | 0 | 1 | 0 | 1

14. Secondary Outcome: Days of Hospitalization
Description: Total number of hospitalization days for hospitalized participants in each group
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Days | 0 (0) | 0 (0) | 6.00 (0) | 0 (0) | 6.00 (0)

15. Secondary Outcome: Cumulative Incidence of Mortality, Measured at Day 28 or Later if Participant is Hospitalized at the Time of Day 28
Time Frame: at Day 28 or later if participant is hospitalized at the time of Day 28 for up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C | Arm D | Arm E
Number analyzed (Participants) | 39 | 39 | 36 | 37 | 35
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 28 and up to 3 months after end of study treatment
Description: Adverse events and serious adverse events were collected from the start of treatment through Day 28 and up to 3 months after the end of the clinical trial. Each event was assessed for severity, seriousness, and relationship to the investigational product.
Groups:
- SOC (Paracetamol): Paracetamol (SOC)
  Standard of care (Paracetamol): SOC - 2 tablets (1000 mg) to be taken 6-hourly as needed
Arm/Group | SOC (Paracetamol) | ASAQ | PA(Pyronaridine-Artesunate) | FPV-NTZ | SOF/DCV
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/39 | 0/38 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/39 | 0/38 | 1/36 | 0/36
Other Adverse Events (participants affected / at risk) | 14/39 | 18/39 | 21/38 | 31/36 | 16/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC (Paracetamol) (N=39) | ASAQ (N=39) | PA(Pyronaridine-Artesunate) (N=38) | FPV-NTZ (N=36) | SOF/DCV (N=36)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SOC (Paracetamol) (N=39) | ASAQ (N=39) | PA(Pyronaridine-Artesunate) (N=38) | FPV-NTZ (N=36) | SOF/DCV (N=36)
nausea (Gastrointestinal disorders) | 2 (2) | 6 (6) | 4 (4) | 8 (8) | 4 (4)
diarrhea (Gastrointestinal disorders) | 5 (5) | 3 (3) | 3 (3) | 7 (7) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 4 (4) | 8 (8) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (5) | 5 (5) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 2 (2) | 9 (9) | 4 (4) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 11 (12) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT04532931/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04532931/SAP_001.pdf